CLINICAL TRIAL: NCT07054775
Title: Comparison of Pruritus Incidence After Intrathecal Morphine 0.1 and 0.2 Milligrams in Cesarean Section: A Randomized Clinical Trial
Brief Title: Comparison of Pruritus Incidence After Intrathecal Morphine 0.1 vs 0.2 mg in Cesarean Section
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Thepakorn Sathitkarnmanee, Associate professor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE631484
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Pruritus Caused by Drug
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Intervention Model Description: Arm 1: intrathecal morphine (ITM) 0.1 mg Arm 2" intrathecal morphine (ITM) 0.2 mg
Who Masked: Participant, Outcomes Assessor
Masking Description: They are unaware of type of drug administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ITM 0.1 mg (Active Comparator): Participants receive spinal anesthesia with 0.5% hyperbaric bupivacaine plus morphine 0.1 mg intrathecally
  Interventions: Drug: Morphine Sulfate
- ITM 0.2 mg (Active Comparator): Participants receive spinal anesthesia with 0.5% hyperbaric bupivacaine plus morphine 0.2 mg intrathecally
  Interventions: Drug: Morphine Sulfate

INTERVENTIONS:
Drug: Morphine Sulfate — intrathecal administered morphine

SUMMARY:
This study compares the incidence of pruritus (itching) requiring treatment between two doses of intrathecal morphine (0.1 mg vs 0.2 mg) when used for spinal anesthesia during cesarean section. The study aims to determine if the lower dose (0.1 mg) can reduce pruritus incidence while maintaining adequate pain relief.

DETAILED DESCRIPTION:
Spinal anesthesia is a standard technique for cesarean section. Intrathecal morphine (ITM) provides prolonged and effective analgesia but may cause adverse events including pruritus, nausea, vomiting, and respiratory depression. Current practice at Srinagarind Hospital uses ITM 0.2 mg for spinal anesthesia in cesarean section. This study investigates whether reducing the ITM dose to 0.1 mg can decrease pruritus incidence while preserving analgesic effectiveness.

ELIGIBILITY:
Inclusion Criteria: • Pregnant women aged 18-45 years

* Full-term pregnancy
* Scheduled for non-emergency cesarean section
* ASA physical status I-III
* Non-complicated pregnancy

Exclusion Criteria:

* Contraindication to spinal anesthesia or study drugs
* Refusal to participate in the study
* BMI ≥ 40 kg/m²
* History of systemic skin disease or current itchy skin condition
* Use of antihistamines or anti-pruritic medications within 3 days prior to surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant female undergoing cesarean section
Enrollment: 69 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of pruritus requiring treatment [Time Frame: 24 hours post-operatively] | 24 hours
  * Percentage of participants requiring treatment for pruritus within 24 hours after spinal anesthesia
  * Measured using numerical rating scale (0-10), with treatment indicated for score ≥4
  * Percentage of participants requiring treatment for pruritus within 24 hours after spinal anesthesia
  * Measured using numerical rating scale (0-10), with treatment indicated for score ≥4
  * Percentage of participants requiring treatment for pruritus within 24 hours after spinal anesthesia
  * Measured using numerical rating scale (0-10), with treatment indicated for score ≥4

CONTACTS AND LOCATIONS:
Overall Officials: Thepakorn Sathitkarnmanee, Study Chair — Faculty of Medicine, Khon Kaen University
Locations (2):
- Thailand (2):
  - Faculty of Medicine, Khon Kaen University, Khon Kaen
  - Thepakorn Sathitkarnmanee, Khon Kaen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kumar K, Singh SI. Neuraxial opioid-induced pruritus: An update. J Anaesthesiol Clin Pharmacol. 2013 Jul;29(3):303-7. doi: 10.4103/0970-9185.117045. PMID 24106351
- [Result] Waxler B, Dadabhoy ZP, Stojiljkovic L, Rabito SF. Primer of postoperative pruritus for anesthesiologists. Anesthesiology. 2005 Jul;103(1):168-78. doi: 10.1097/00000542-200507000-00025. PMID 15983470
- [Result] Sultan P, Halpern SH, Pushpanathan E, Patel S, Carvalho B. The Effect of Intrathecal Morphine Dose on Outcomes After Elective Cesarean Delivery: A Meta-Analysis. Anesth Analg. 2016 Jul;123(1):154-64. doi: 10.1213/ANE.0000000000001255. PMID 27089000
- [Result] Gehling M, Tryba M. Risks and side-effects of intrathecal morphine combined with spinal anaesthesia: a meta-analysis. Anaesthesia. 2009 Jun;64(6):643-51. doi: 10.1111/j.1365-2044.2008.05817.x. PMID 19462494
- [Result] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Result] Wang W, Zhou L, Sun L. Ondansetron for neuraxial morphine-induced pruritus: A meta-analysis of randomized controlled trials. J Clin Pharm Ther. 2017 Aug;42(4):383-393. doi: 10.1111/jcpt.12539. Epub 2017 May 2. PMID 28464238